CLINICAL TRIAL: NCT05389943
Title: The Effect of Vitamin D3 Therapy in Post Menopausal Women and Assessment of Changes in Bone Mineral Density
Brief Title: The Effect of Vitamin D3 Therapy in Post Menopausal Women and Assessment of Changes in Bone Mineral Density After Orally Vitamin D3 Administration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sargodha (Other)
Collaborators: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Muhammad irsalan, Medical officer, University of Sargodha
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: USargodha
Record Dates: First submitted 2022-05-21; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Vitamin D Deficiency
Keywords: Postmenopausal women, Low Bone density
MeSH Terms: conditions — Vitamin D Deficiency; Bone Diseases, Metabolic | interventions — Milk; Diet

STUDY DESIGN:
Intervention Model Description: Randomized control trial on OPD patients (female age above 50) postmenopausal. the effect of vitamin D supplement on these women's bone density.
Who Masked: Participant, Care Provider
Masking Description: participants and care giver will be blind in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Postmenopausal women with low BMD (Experimental): patient with serum 25-hydroxy vitamin D [25(OH)D] less than 32 ng/ml. Vitamin D3 5000 IU/d per oral for the period of 3 months will be administered
  Interventions: Drug: Oral administration of vitamin D3; Drug: Vitamin D3 50000 UNT Oral Capsule; Dietary Supplement: milk, Dietary and life style modifications.
- Postmenopausal women (Active Comparator): Postmenopausal women having serum 25-hydroxy vitamin D [25(OH)D] greater than 32 ng/ml will provided with milk and dietary modifications.
  Interventions: Dietary Supplement: milk, Dietary and life style modifications.

INTERVENTIONS:
Drug: Oral administration of vitamin D3 — the effect of oral supplement in postmenopausal women.
  Other Names: Postmenopausal women
  Arms: Postmenopausal women with low BMD
Drug: Vitamin D3 50000 UNT Oral Capsule — In postmenopausal women with BMD less than 32 ng/ml
  Arms: Postmenopausal women with low BMD
Dietary Supplement: milk, Dietary and life style modifications. — Postmenopausal women with BMD greater than 32 ng/ml

SUMMARY:
a study design based on vitamin D deficiency in postmenopausal women with low bone density. pre-test for BMD will be done then vitamin D oral supplements will be provided for the period of 3 months. Post-test of BMD will explore the results.

DETAILED DESCRIPTION:
Sample description Study Design Randomized Control Trial. Settings OPD patients Duration 8 months Sample size 200 Masking Single blind (only Participants) Study subjects Routine visit OPD patients with orthopedic problems Sampling techniques RCT will be done by giving vitamin D (pre-test and post-test of BMD will be done .

Inclusion Criteria Female patients above 50 years (Post-menopausal) Exclusion Criteria All other women Study variables : Independent: Vitamin D Data collection will be done through randomized control trial. Patient with age above 50 years female, with menopausal changes. The BMD test will be done in all participants either placebo or actual treated patients to check the effect of vitamin D3 therapy. Treatment plan includes vitamin D3 at 50,000 International Units daily for 15 days then two times a month for four months along with dietary changes which will consider high dose D3 therapy, and low dose vitamin D3 therapy includes dietary changes along with 1000 international units of Vitamin D3 tablet form. Daily white placebo pills to other group of participants. Bone Mineral Density will be observed through pre-test and Post-test.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Women

Exclusion Criteria:

* All other women

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — More than 50 years old
Enrollment: 80 (Estimated)
Dates: Start 2022-06-05 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Postmenopausal women BMD will be improved with oral vitamin D supplements | 3 to 4 months
  Vitamin D can improve the BMD in women and reduces the risk of infection

CONTACTS AND LOCATIONS:
Locations (1):
- Arsalan Khalid, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
not decided yet